CLINICAL TRIAL: NCT04677998
Title: A Personalized Surveillance and Intervention Protocol for Duodenal and Gastric Polyposis in Patients With Familial Adenomatous Polyposis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Leiden University Medical Center (Other); The Netherlands Cancer Institute (Other); St Mark's Hospital Foundation (Other); Hospital Clinic of Barcelona (Other); Hôpital Edouard Herriot (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Hospital General Universitario de Alicante (Other); University Medical Center Mainz (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Prof. Evelien Dekker, MD, PhD, Prof. dr. Evelien Dekker, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W20_181
Record Dates: First submitted 2020-11-24; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Endoscopic surveillance; Endoscopic interventions; Personalized care; Gastrointestinal neoplasia
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Personalized surveillance and intervention protocol
  Interventions: Procedure: Personalized surveillance and intervention protocol

INTERVENTIONS:
Procedure: Personalized surveillance and intervention protocol — This study uses one arm. Participants will undergo endoscopic surveillance with intervals between 3-6 months and 5 years, depending on severity of polyposis and performed endoscopic interventions.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a personalized surveillance and intervention protocol for duodenal and gastric polyposis in patients with familial adenomatous polyposis (FAP)

DETAILED DESCRIPTION:
Patients with FAP are not only at risk of developing colorectal adenomas but also at high risk of developing duodenal adenomas. In 30% to 92% of FAP patients duodenal adenomas are detected, with a lifetime risk approaching 100%. Of these duodenal adenomas, only a small proportion develops into duodenal cancer, with a prevalence of approximately 5-10% in FAP patients.

Endoscopic surveillance is nowadays the standard of care to prevent FAP patients from developing duodenal cancer. The severity of duodenal polyposis is assessed using the Spigelman classification system. This classification is based on the number, size, histology, and grade of dysplasia of the duodenal adenomas, resulting in a score varying from 0-IV, guiding surveillance intervals and treatment.

Concerns are rising on the accuracy of the Spigelman score as predictor for duodenal cancer, especially for ampullary cancer. Over the past years, multiple studies demonstrated limitations of this staging system including the fact that this classification does not adequately predict duodenal/ampullary cancer and does not guide endoscopic or surgical interventions. A clear endoscopic intervention protocol is needed, not only to prevent the development of cancer but also to prevent the need for duodenal surgery, since these surgical procedures are associated with high complication and mortality rates.

With this study, the investigators aim to evaluate a personalized surveillance and intervention protocol for the duodenum and stomach with the goal to prevent the development of advanced neoplasia (AN) by endoscopically removing lesions before they progress to AN.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FAP, at least one of following: genetic diagnosis (proven APC germline mutation) and/or clinical diagnosis (>100 colorectal adenomas in combination with a positive family history of FAP)
* Age 18 years or older

Exclusion Criteria:

* Endoscopic removal of all polyps with an indication for removal not possible/feasible
* Gastric or duodenal cancer at baseline endoscopy
* Need for surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with FAP treated at one of the participating centers will be assessed for eligibility.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Advanced neoplasia | Up to 5 years
  Incidence of advanced neoplasia defined as adenomas ≥15mm, high grade dysplasia (HGD) and/or duodenal/ampullary cancer

SECONDARY OUTCOMES:
Recurrences after different endoscopic intervention techniques | Analysis at 2 years and 5 years
  Incidence of recurrences after endoscopic interventions after en bloc/piecemeal resection and different techniques such as cold snare polypectomy or endoscopic mucosal resection with or without lifting
Feasibility of endoscopic interventions | Analysis at 2 years and 5 years
  Incidence of lesions not amenable to endoscopic removal
Accuracy optical diagnosis | Analysis at 2 years and 5 years
  The ability of endoscopists to optically diagnose duodenal and gastric lesions. Sensitivity and specificity for optically diagnose high-grade dysplasia in the stomach and duodenum.
Complications | Analysis at 2 years and 5 years
  Incidence of endoscopy related complications
Surveillance burden | Up to 5 years
  Surveillance burden (number of endoscopies for each patient)
Surgery | Up to 5 years
  Incidence of surgical interventions

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, North Holland, Netherlands